CLINICAL TRIAL: NCT03041350
Title: Smartphone Video-assisted Advanced Life Support of Patients With Out-of-hospital Cardiac Arrest by EMS Under Physician Direction
Acronym: SWALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Public Safety and Security (Unknown); Ajou University School of Medicine (Other); Saint Vincent's Hospital, Korea (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Yu Jin Kim, MD, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SWALS
Record Dates: First submitted 2016-12-11; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Emergency Medical Services; Smartphone; Survival
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

ARMS (1):
- Smartphone video-assisted ALS & Conventional CPR (Experimental): In study period, using this video medical control, high-quality CPR, cardiac arrest rhythm confirmation, defibrillation, proper drug administration instructions, advanced airway insertion, etc. are performed. The medical director then decides on patient transfer if the asystole and pulseless electrical activity findings are persistent even after more than 20-minutes of ALS.
  The conventional CPR is Basic life support only in the automatic external defibrillator (AED) mode 5-10 minutes at the scene, are not allowed to stop resuscitation at the scene unless there is a return of spontaneous circulation (ROSC) or pre-hospital cardiac arrest patient has already been transported to a hospital.
  Interventions: Other: Smartphone video-assisted ALS(advanced life support)

INTERVENTIONS:
Other: Smartphone video-assisted ALS(advanced life support) — As an preparation for this study, personnel training in mock advanced life support (ALS) simulation including the smartphone video call methodology was conducted. The smartphones were not separately purchased or produced; commercially available smartphones already owned by the emergency medical service (EMS) personnel and medical directors were used. To facilitate the smartphone video call between the medical director and the EMS personnel and to prevent the caregivers or others nearby from hearing the conversation, Bluetooth earphone sets were used. Data were collected using the cardiopulmonary resuscitation (CPR) recording form uploaded in SNS which consisted of EMS personnel and medical directors, and the quality of CPR was evaluated

SUMMARY:
Direct medical control using video conferencing capabilities of smartphones has never been conducted in out-of-hospital cardiac arrest patients. This study was conducted to investigate its feasibility and treatment effectiveness in out-of-hospital cardiac arrest (OHCA) patients using a real-time smartphone video call.

DETAILED DESCRIPTION:
If cardiac arrest is suspected, the EMS personnel contacted the medical director before arriving at the scene. Upon the arrival at the scene of the two activated paramedic teams, they rapidly switch to ALS under teamwork-based BLS and video medical control. Using this video medical control, high-quality CPR, cardiac arrest rhythm confirmation, defibrillation, proper drug administration instructions, advanced airway insertion, etc. are performed. The medical director then decides on patient transfer if the asystole and pulseless electrical activity findings are persistent even after more than 20-minutes of ALS. After initiating the transfer, the medical director contacts the hospital where the patient is to be transferred to after completing the video medical control. The medical director provides an explanation of the treatment to the caregiver via video. After returning to the fire station, the EMS personnel who had completed the patient's transfer the enters the information by hand on the separate form, takes a picture of the document, and uploads it to SNS within 24 hours. Through this information shared via SNS, the research staff the provides a direct feedback to the EMS personnel, and further discussion performed within the SNS. All the incident cases of OHCA during the before and during interventional periods were registered using an EMS run sheet for basic ambulance operation information, the EMS cardiac arrest registry for the Utstein factors, and the OHCA registry for the hospital care and survival outcomes. The EMS run sheet and EMS cardiac arrest registry were collected by the EMS providers. The medical records for hospital care and outcomes were abstracted by the trained reviewer for this study

ELIGIBILITY:
Inclusion Criteria:

* all EMS-treated OHCA patients older than 18 years transported to the hospital unless otherwise diagnosed with trauma, poisoning, asphyxia, hanging, or any other non-disease-origin factors.

Exclusion Criteria:

* Patients with do-not-resuscitate (DNR) orders and with obvious signs of irreversible death, including rigor mortis and corruption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
survival rate | 1 year
favorable neurologic outcome rate | 1 year

SECONDARY OUTCOMES:
rate of prehospital return of systemic circulation(ROSC) | through study completion, an average of 1 year

OTHER OUTCOMES:
feasibility | through study completion, an average of 1 year
  Confidence scores of 10 items for determining CPR performances which is measured on a 10 point likert scale by physicians

CONTACTS AND LOCATIONS:
Overall Officials: Gi Woon Kim, M.D., Ph.D., Principal Investigator — Department of Emergency Medicine, Soonchunhyang University Bucheon Hospital
Locations (1):
- Emergency medical service system of Suwon city, Suwon, Gyeonggi-do, South Korea